CLINICAL TRIAL: NCT02892643
Title: Multicenter Prospective Randomized Controlled Trial of Comparing Laparoscopic Proximal Gastrectomy and Laparoscopic Total Gastrectomy for Upper Third Early Gastric Cancer (KLASS-05)
Brief Title: Comparison of Laparoscopic Proximal Gastrectomy and Laparoscopic Total Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Do Joong Park, M.D., Ph.D., Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1609-361-001
Record Dates: First submitted 2016-09-02; First posted 2016-09-08 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Laparoscopic proximal gastrectomy (Experimental): Laparoscopy proximal gastrectomy with esophago-jejunostomy, gastro-jejunostomy and jejuno-jejunostomy (double tract reconstruction). Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.
  Interventions: Procedure: Laparoscopic proximal gastrectomy
- Laparoscopic total gastrectomy (Active Comparator): Laparoscopic total gastrectomy with esophago-jejunostomy and jejuno-jejunostomy (Roux-en-Y reconstruction). Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.
  Interventions: Procedure: Laparoscopic total gastrectomy

INTERVENTIONS:
Procedure: Laparoscopic proximal gastrectomy — Laparoscopy proximal gastrectomy with esophago-jejunostomy, gastro-jejunostomy and jejuno-jejunostomy (double tract reconstruction). Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.
  Arms: Laparoscopic proximal gastrectomy
Procedure: Laparoscopic total gastrectomy — Laparoscopic total gastrectomy with esophago-jejunostomy and jejuno-jejunostomy (Roux-en-Y reconstruction). Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.
  Arms: Laparoscopic total gastrectomy

SUMMARY:
Experimental: Laparoscopic proximal gastrectomy Laparoscopy proximal gastrectomy with esophago-jejunostomy, gastro-jejunostomy and jejuno-jejunostomy (double tract reconstruction). Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.

Active Comparator: Laparoscopic total gastrectomy Laparoscopic total gastrectomy with esophago-jejunostomy and jejuno-jejunostomy (Roux-en-Y reconstruction). Systemic en bloc lymph node dissection is mandatory. Resection margin should be negative for malignancy with intraoperative frozen biopsy.

DETAILED DESCRIPTION:
Participating Surgeons Prior to this clinical trial, only the surgeons who are considered to have the standardization by review committee participated.

Patients Registration It is required to ensure that the patients meet the inclusion criteria for this clinical trial, are free from any items of exclusion criteria, are explained about the participation in the clinical trial along with the informed consent forms.

After rechecking the patients with the registration check list by accessing the web-based randomized program provided from Seoul National University Bundang Hospital Medical Research Collaborating Center.

Each group 69 patients, total 138 subjects will be enrolled. Randomization The registration randomization should be done with 1:1 ratio for each researcher.

Baseline number (BN) should be provided to the subjects in the order of acquisition of informed consent form. Based on the subjects who are selected as the appropriate subjects in the end, the allocation number (AN) shall be provided in the order of randomized allocation table.

Procedure Operations are performed according to the allocated group.

ELIGIBILITY:
Inclusion Criteria:

* Patients are included in the trial if they meet all of the following criteria:

Histologically proven adenocarcinoma through endoscopic biopsy Aged 20-80 years old Written signed informed consent No other malignancies Proximal gastric cancer met by following conditions ; Lesion located on proximal stomach (upper one third) Lesion below 5cm in size Lesion confined to mucosa or submucosa (cT1) No evidence of metastatic enlarged LN on #5, 6, 4d, 10 basins and other distant metastasis.

Performance status (PS) of 0 or 1 on Eastern Cooperative Oncology Group (ECOG) scale Performance status (PS) of I to III on American Society of Anesthesiologists (ASA) score

Exclusion Criteria:

* Patients are excluded if they meet any of the following criteria:

History of anemia Patients who need total gastrectomy History of pre-operative chemotherapy or radiation therapy for gastric cancer Patients who need combined resection (except cholecystectomy) Presence of other malignancies Prior treatment against systemic inflammatory disease Previous gastric surgery Vulnerable patients (lack of decision-making capacity, pregnant, or breast-feeding women)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-10-27; Primary Completion 2018-09-17 (Actual); Study Completion 2020-09-17 (Actual)

PRIMARY OUTCOMES:
Change of Hemoglobin | up to 2 years postoperatively
  from blood sample
Vitamin B12 cumulative supplement quantity | up to 2 years postoperatively
  from blood sample

SECONDARY OUTCOMES:
Operative morbidity | 30 days for early morbidity
  Complications occuring after operation
Operative mortality | mortality for 90 days
  Mortality after operation
QOL measurement | 6 month, 1 year, 2 year, postoperatively
  EORTC C30/STO22
Reflux esophagitis | check at every 12 months up to 2 years postoperatively
  assessed by Visick score and endoscopic grading according to LA classification
Relapse-free survival | 2 years postoperatively
  Relapse-free survival
Overall survival | 2 years postoperatively
  Overall survival

CONTACTS AND LOCATIONS:
Locations (16):
- South Korea (16):
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - Dong-A University Hospital, Busan
  - Dankook University Hospital, Cheonan
  - Keimyung University Hospital, Daegu
  - Chungnam National University Hospital, Daejeon
  - Eulji University Hospital, Deajon, Daejeon
  - Chonnam National University Hospital, Hwasun
  - National Cancer Center, Ilsan
  - Pusan National University Hospital, Pusan
  - Seoul National University Bundang Hospital, Seongnam
  - Ewha Womans University Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul St. Mary's Hospital, Seoul
  - Yeouido St. Mary's Hospital, Seoul
  - Yonsei University Severance Hospital, Seoul
  - Ajou University Hospital, Suwon

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park DJ, Han SU, Hyung WJ, Hwang SH, Hur H, Yang HK, Lee HJ, Kim HI, Kong SH, Kim YW, Lee HH, Kim BS, Park YK, Lee YJ, Ahn SH, Lee I, Suh YS, Park JH, Ahn S, Park YS, Kim HH. Effect of Laparoscopic Proximal Gastrectomy With Double-Tract Reconstruction vs Total Gastrectomy on Hemoglobin Level and Vitamin B12 Supplementation in Upper-Third Early Gastric Cancer: A Randomized Clinical Trial. JAMA Netw Open. 2023 Feb 1;6(2):e2256004. doi: 10.1001/jamanetworkopen.2022.56004. PMID 36790808
- [Derived] Hwang SH, Park DJ, Kim HH, Hyung WJ, Hur H, Yang HK, Lee HJ, Kim HI, Kong SH, Kim YW, Lee HH, Kim BS, Park YK, Lee YJ, Ahn SH, Lee IS, Suh YS, Park JH, Ahn S, Han SU. Short-Term Outcomes of Laparoscopic Proximal Gastrectomy With Double-Tract Reconstruction Versus Laparoscopic Total Gastrectomy for Upper Early Gastric Cancer: A KLASS 05 Randomized Clinical Trial. J Gastric Cancer. 2022 Apr;22(2):94-106. doi: 10.5230/jgc.2022.22.e8. PMID 35534447